CLINICAL TRIAL: NCT04219124
Title: The Effect of a SGLT2 Inhibitor on Glucose Flux, Lipolysis and Exercise in Type 2 Diabetes
Acronym: SINGLED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: Royal Surrey County Hospital NHS Foundation Trust (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 0585
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin

STUDY DESIGN:
Intervention Model Description: The study is a randomised double blind placebo control cross over trial. with 4-weeks washout period.
Who Masked: Participant, Investigator
Masking Description: Matching placebo for Dapagliflozin 10 mg. Dosage form and strength: Green, plain, diamond shaped, and film coated tablet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Active Comparator): Investigational product: Dapagliflozin 10 mg Dosage form and strength: Green, plain, diamond shaped, film coated 10 mg tablet with frequency of 1 tablet per day for 4 weeks
  Interventions: Drug: IMP oral tablet
- Placebo (Placebo Comparator): Investigational product: Matching placebo for Dapagliflozin 10 mg. Dosage form and strength: Green, plain, diamond shaped, and film coated tablet with frequency of 1 tablet per day for 4 weeks
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: IMP oral tablet — Dapagliflozin 10 MG
  Other Names: Farexiga, gliflozin class, SGLT2 inhibitor
  Arms: Dapagliflozin
Drug: Placebo oral tablet — Matching placebo tablets
  Other Names: Matching placebo tablet for dapagliflozin 10 MG
  Arms: Placebo

SUMMARY:
The study is a randomised double blind placebo control cross over trial with 4 weeks washout period. The expected duration of participant participation is 103 days. the study aims to investigate the effect of dapagliflozin, a SGLT2 inhibitor, on glucose flux, lipolysis and exercise in patients with type 2 diabetes.

DETAILED DESCRIPTION:
SGLT2 inhibitors are a new class of drug that have a novel mechanism of action by promoting urinary glucose excretion to lower blood glucose levels. The recent observations that ketogenesis or episodes of diabetic ketoacidosis seem to be of higher frequency in patients with Type 1 and Type 2 diabetes on SGLT2 inhibitors, is of considerable worldwide interest. SGLT2 inhibitors seem to be associated with euglycemic DKA and ketosis, perhaps because of their noninsulin-dependent glucose clearance, hyperglucagonemia, and volume depletion. There have been two papers that have looked at this in some detail. One is a metabolic study by Ferrannini et al and a review paper by Yabe et al. The central question that needs to be raised is whether the observed effects are solely due to the SGLT2 inhibitors masking elevations in blood glucose in insulin deficient states, or whether there is some metabolic effect of the SGLT2 inhibitors that make episodes more likely to occur. There is increasing evidence to suggest that the SGLT2 inhibitors are affecting metabolism in several ways and that these may contribute to the risk of ketoacidosis. Ferrannini et al have shown that, on chronic usage, lipid oxidation rates change and thus the body appears to have a homeostatic response to losing glucose by switching metabolism more in favour of free fatty acids. It is also possible that protein and other metabolites are also involved in this process but these have never been studied.

Recent trials of newer glucose-lowering agents have been neutral on the primary Cardiovascular (CV) outcome. However, patients with type 2 diabetes at high risk for cardiovascular events who received empagliflozin, as compared with placebo, had a lower rate of the primary composite cardiovascular outcome and of death from any cause when the study drug was added to standard care. This may be a class effect and is of high importance to explore the effects of SGLT2 inhibitor effect on cardiovascular function.

Aim: To study the metabolic adaptions that take place following chronic administration of SGLT2 inhibitors in people with Type 2 diabetes and to establish whether these adaptations contribute to the development of ketoacidosis.

Study procedure:

The recruitment phase will commence as soon as there is ethical, HRA, research governance and regulatory approval and only after the Sponsor 'green light' has been issued.

Recruitment: From Diabetes Clinics at Cedar centre, Royal Surrey County Hospital and additional locations: local GP practices, other healthcare settings including but not limited to outpatient clinics, retinal screening, podiatry, diabetes patient groups, University of Surrey staff.

Participants will be screened by the diabetes research team, which includes research doctors and nurses working at the Cedar centre research unit.

Informed Consent- The participant will have a minimum of 24hours to consider participation in the study to consider the information, and the opportunity to question the Investigator, their GP or other independent parties to decide whether to participate in the study. Written Informed Consent will then be obtained.

If the individual fulfils the inclusion criteria and meets none of the exclusion criteria they will be accepted into the study. All females of childbearing age will need to provide a urine sample for a pregnancy test.

Diastolic blood pressure, systolic blood pressure, and pulse will be taken in line with the Cedar centre SOP. Any abnormal or clinically significant deterioration will be reported as an adverse event.

Weight and height will be recorded at screening visit and weight only at visits 2- 6. Weight (without shoes) will be measured using body composition analyser. Height (without shoes) recorded using a stand-alone stadiometer for height measurement, manufacturer unknown. Body Mass Index (BMI) will be calculated and rounded up/down to nearest whole figure at each visit.

Physical examination will be carried out. Any abnormal, clinically significant findings at screening visit must be recorded as concomitant illness.

If acute kidney injury occurs, the study medication will be promptly discontinued and kidney impairment treated using standard guidelines.

Laboratory Tests Point of care or plasma HbA1C within 1 month of the screening visit. All laboratory results will be reviewed, and the reports signed by the Investigator or delegate in accordance with the delegation log, who will record in the CRF whether they are normal, abnormal but not clinically significant, or abnormal and clinically significant. In the latter case the eligibility of the participants will be reviewed.

Bloods samples analysed at University of Surrey will be viewed as bloods of research significance and not reported to the GP.

Subsequent Assessments:

Visit 2: week 1: Baseline VO2 max test A VO2 max test will be used to tailor exercise intensity to each participant. This exercise intensity information will be used for visit 3 and 5 when the exercise test is completed.

Participants will use an exercise bike and wear a mask and mouthpiece. Participants will perform a 5min warm up at 25% VO2 max. The submaximal exercise test using a 2-stage bicycle ergometer protocol will consist of two consecutive 10min stages at a constant load corresponding to 40 and 70 % VO2 max followed by 5 min warm down. In addition, measurements relating to heart function will be taken.

Visit 3 and 5: Exercise test Participants will have a standardised meal the evening before the exercise test and will arrive at the laboratory after an overnight fast. The standardised meal is 500-kcal meal, which will be provided by the study team for the participant to prepare and cook at home.

A cannula will be inserted into an antecubital vein and baseline blood samples taken at times 0, 5, 10, 15, 20, 25, 30 and 60 min before, during and after exercise.

Participants will be asked to complete a set duration of exercise on the exercise bike. The duration and intensity will have been calculated from the results of visit 2. They will wear a mouthpiece and mask throughout and be attached to a cardiac monitor.

The following measurements will be taken before and during/after exercise:

* Plasma non-esterified fatty acid concentrations, atrial natriuretic peptide, noradrenaline and adrenaline (n=8 for each measurement)
* Plasma glucose, insulin and growth hormone concentrations (n=8 for each measurement)
* Ketone body and metabolite concentrations (n=8 for each measurement)
* ECG trace
* BP, HR and Rate Pressure Product (RPP=HR*SBP)
* Calculated substrate oxidation recorded as VO2 ml/min and VCO2 ml/min and resting energy requirement (RER)
* Capillary lactate concentration Visit 4 and 6: The Metabolic Assessment Day (8-10 hours) Participants will have taken the randomised study treatment daily for 28 days prior to visit 4 and 6. Blood glucose study diaries will be collected at visit 4 and 6. Hypoglycaemia events will be reviewed. Data from their home glucose monitoring will not be collected for further analysis.

Participants should refrain from alcohol and strenuous exercise for 24hours prior to any metabolic assessment day. If female of childbearing age, a urine pregnancy test will be undertaken prior to the commencement of any metabolic study activity. Blood pressure and heart rate will be recorded. Participants will be asked to return their unused IMP at visit 4 and visit 6. They will be prescribed the IMP required for the second arm of the study depending on the randomisation code.

Participants will have a standardised meal the evening before the metabolic assessment day and will attend the clinical research unit at 7.00am on the morning of the assessment day after an overnight fast. Blood glucose concentration will be measured using a glucose oxidase technique on a glucose analyser (YSI 2300 Clandon Scientific, Yellow Springs Instruments, Yellow Springs, Ohio, USA). Hydration may be maintained by insertion of an intravenous fluid drip.

All blood samples will be separated immediately using a centrifuge (Heraeus Labofuge 400 centrifuge, Thermo Fisher Scientific. UK) and the plasma stored at -20°c at the Cedar centre overnight and then transferred to a minus -80°c freezer at the University of Surrey for analysis later at the University of Surrey.

Metabolic Assessment Day Blood samples will be as shown in Appendix A. The samples will be used for measuring different metabolites and hormones at various time points.

Intravenous cannulae will be inserted into the antecubital fossa of each arm: one for blood taking at time -15 minutes and the other for the infusion of the isotopes [6,6]- 2H2 glucose and [1,1,2,3,3]- 2H5 glycerol at time 360 minutes. Two fasting samples will be taken at -10 and 0 for the baseline isotope enrichment for glucose, glycerol and palmitate and NEFA and ketone body concentrations and various hormone concentrations.

At 0 minutes the study medication will be taken and a stable isotope of U-13C palmitate (200mg) in 30 ml olive oil will be ingested in less than 2 minutes after which blood samples will be taken for palmitate enrichment and concentration in TAG and NEFA pools and TAG and NEFA concentrations.

A primed infusion of stable isotope of glucose and glycerol will be given from 360 to 480 minutes and the concentration and enrichment of both glucose and glycerol will be measured from 450 minutes to 480 minutes.

Samples will be taken for glucose concentration throughout the study. Blood samples for acetoacetate concentration and beta-hydroxybutyrate enrichment and concentration will be taken.

One blood sample will be taken at 480 minutes for targeted metabolomics and cardiac biomarkers.

Blood samples for will also be taken for insulin, glucagon and cortisol. Patients will be asked to empty their bladder and urine will be collected to analyse glucose excretion at 120, 360, 450 and 480 minutes (4 samples).

A Transthoracic Echocardiogram and pulse wave velocity will be completed during the metabolic assessment day. This can be done at any time point during the metabolic assessment day.

On completion of the metabolic assessment day, participants will be reminded that they have the telephone number for the research team that can be used 24hours a day (identification card) and will be advised not to drive home.

There will be a minimum period of a 28-day drug wash out period before starting the second arm of the study. The participant will be dispensed with trial medication for the second arm at visit 4. A date will be agreed for visit 5 and 6 to allow the study doctor to advise when the participant should to start taking the study medication in preparation for visit 5 and 6.

Telephone Visits 1 and 2 The research team will contact the participant the day after each metabolic assessment day to ensure glucose levels have normalised. This may be a Saturday if a metabolic study is conducted on a Friday.

Telephone Visit 3 Once participants have completed both metabolic assessments days the participant will have completed the research study protocol. Each participant will receive a follow up check on well-being 2-4 weeks after completion of the last metabolic assessment day and will continue their diabetes care with their usual diabetes doctor.

If a participant withdraws from the study, all samples will be destroyed but the anonymised data collected up to the point of withdrawal will be used unless explicitly stated by the participant. The study doctor may also decide that it is no longer appropriate for a participant to continue with the study. This will happen if they no longer meet the requirements for the study or exclusion criteria become apparent. The participant will be required to withdraw from the study if they become pregnant or lose capacity to follow the study procedures and provide consent to continue.

ELIGIBILITY:
Inclusion Criteria:

* • Able in the opinion of the investigator, and willing to give informed consent obtained before any study-related activities.

  * Diagnosis of type 2 diabetes greater than 12 months.
  * Single, dual or triple therapy glucose lowering agents comprising of sulphonylureas, biguanides and DDP-IV.
  * No previous exposure to SGLT2 inhibitors.
  * BMI of less than 40.
  * HbA1c of greater or equal to 6.5% and less than 9% within 1 month of screening.
  * Able to comply with the study and the study procedures.
  * Patients who are or who have previously been involved in research are eligible provided a participant has not received an investigational drug within one month of entry into the study.

Exclusion Criteria:

* • Participants over 75.

  * Participants under 18.
  * Participants who cannot adequately understand verbal and / or written explanations given in English.
  * Clinical suspicion of Hypoglycaemic unawareness.
  * LADA -latent autoimmune diabetes in adults due to differing nature of the illness/Type 1.
  * Confirmed excessive and compulsive drinking of alcohol i.e. alcohol abuse as determined from GP medical notes by the Fast Alcohol Screening Test (FAST) or history of previous alcohol abuse.
  * Has a history of chronic pancreatitis.
  * Restricted food intake - Determined by history.
  * Diagnosis of osteoporosis confirmed by DEXA scan.
  * Participants on insulin, insulin analogs or GLP-1 in the preceding 6 months.
  * Proliferative retinopathy that has required acute treatment within last three months.
  * Moderate to severe renal impairment (creatinine clearance [CrCl] < 60 ml/min or estimated glomerular filtration rate [eGFR] < 60 ml/min/1.73 m2.
  * History of unstable or rapidly progressing renal disease.
  * Severe hepatic insufficiency / and or significant abnormal liver function defines as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and / or alanine aminotransferase (ALT) > 3ULN.
  * Positive serologic evidence of current infectious liver disease including Hepatitis B viral antibody IGM, Hepatitis B surface antigen and Hepatitis C virus antibody.
  * Congestive heart failure defined as New York Heart Association (NYHA) class III and IV, unstable or acute congestive heart failure.
  * Uncontrolled cardiac arrhythmias.
  * Uncontrolled hypertension. (BP greater than 160/90).
  * Mental incapacity.
  * Pregnancy or breast feeding women.
  * Those of child-bearing potential not taking adequate contraception precautions. Adequate protection is defined as barrier protection, oral contraceptive pill or intrauterine device.
  * Volume depleted patients, patients at risk of volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics should have careful monitoring of their volume status.
  * History of unstable angina.
  * Acute Coronary Syndrome (ACS) within 2 months prior to enrolmen.t
  * Hospitalisation for unstable angina or acute myocardial infarction within 2 months prior to enrolment.
  * Acute Stroke or TIA within two months prior to enrolment.
  * Less than two months post coronary artery revascularisation.
  * History of diabetic ketoacidosis (DKA) requiring medical intervention (e.g. emergency room visit and/or hospitalisation) within 1 month prior to the screening visit.
  * Known or suspected allergy to study products.
  * Known Lactose-intolerant.
  * Have severe and enduring mental health problems.
  * Are not primarily responsible for their own care

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of 3-hydroxybutyrate | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 4 and visit 6, concentration of 3-hydroxybutyrate in plasma at baseline and during the visit (hourly for 8hr) will be measured by an enzymatic assay using PENTRA clinical chemistry analyser. The mean concentration of 3-hydroxybutyrate between 420-480 mins and the AUC of 3-hydroxybutyrate concentration time curve between 0-240 mins and 0-480 mins where the IMP was given at 0 mins in visits 4 and 6 will be calculated.The response will be compared following 4 weeks treatment with dapagliflozin versus placebo.

SECONDARY OUTCOMES:
Response to exercise testing: Plasma non-esterified fatty acid (NEFA) concentrations | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 3 and visit 5, plasma NEFA concentrations will be measured by an enzymatic assay using a clinical chemistry analyser (PENTRA). Plasma NEFA concentration measured at 0 minutes and at the end of each level of activity and AUC (0-60 minutes) and will be compared following 4-weeks dapagliflozin versus placebo treatment.
Response to exercise testing: Plasma 3-hydroxybutyrate (BOHB) concentration | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 3 and visit 5, plasma BOHB concentrations will be measured by an enzymatic assay using a clinical chemistry analyser (PENTRA). Plasma BOHB concentration measured at 0 minutes and at the end of each level of activity and AUC (0-60 minutes) and will be compared following 4-weeks dapagliflozin versus placebo treatment.
Response to exercise testing: Atrial natriuretic peptide, noradrenaline and adrenaline | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 3 and visit 5, plasma ANP, noradrenaline and adrenaline measured by ELISA assays. Atrial natriuretic peptide, noradrenaline and adrenaline concentrations will be measured at 0 minutes and at the end of each level of activity and AUC (0-60 minutes) will be compared following 4-weeks dapagliflozin versus placebo treatment.
Response to exercise testing: Glucose concentration, insulin and growth hormone | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 3 and visit 5, plasma glucose concentration measured by an enzymatic assay on PENTRA, a clinical chemistry analyser and insulin and GH concentrations measured by respective radioimmune assays (RIA). Plasma glucose, insulin and growth hormone concentrations will be measured at 0 minutes and at the end of each level of activity and AUC (0-60 minutes) and AUC (0-60 minutes)will be compared following 4-weeks dapagliflozin versus placebo treatment.
Response to exercise testing:ECG abnormality | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 3 and visit 5, ECG taken at rest and during exercise will be compared following 4-weeks dapagliflozin versus placebo
Response to exercise testing: BP, HR and Rate Pressure Product (RPP=HR*SBP) | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 3 and visit 5, blood pressure (BP) and heart rate taken at rest and during exercise. BP, HR and Rate Pressure Product (RPP=HR*SBP) will be measured at 0 minutes and at the end of each level of activity will be compared following 4-weeks dapagliflozin versus placebo
Response to exercise testing: Carbohydrate and fat oxidation | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 3 and visit 5, volumes of inhaled and expired air measured by a Cardio2 Med Graphics breath analyser, (VO2 and VCO2) taken at rest and at the end of each level of activity will allow calculation of carbohydrate and fat oxidation using established mathematical formula. These will be compared following 4-weeks dapagliflozin versus placebo
Response to exercise testing: whole blood capillary lactate concentration | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 3 and visit 5, whole blood capillary lactate concentration measured by single use test strips (lactate Pro) containing an enzyme coated electrode using a lactate analyser (Lactate Pro) in response to exercise at the end of each exercise activity level will be analysed following 4 weeks treatment with dapagliflozin versus Placebo.
Endogenous glucose production and glucose metabolic clearance rate | The main analysis will be conducted once all participants have completed the metabolic studies approximately within 2 years
  At visit 4 and visit 6, plasma glucose enrichment will be measured at basal and in in the last 30 minutes of 2H2-glucose infusion (450-480 min). Enrichment of 2H2glucose in plasma glucose will be measured using gas chromatography mass spectroscopy. Glucose production rate and MCR will be calculated from glucose enrichment data using standard isotope dilution equations. Glucose uptake will be determined by subtracting the rate of glucose excretion from the rate of glucose disappearance. Glucose concentration will be measured as AUC (0-240 minutes), AUC (0-360 minutes), AUC (0-480 minutes)
Glycerol production rate | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 4 and visit 6, plasma glycerol enrichment will be measured at basal and in in the last 30 minutes of 2H5-glycerol infusion (450-480 min). Glycerol production rate and MCR will be calculated from glycerol enrichment data using standard isotope dilution equations.
Palmitate enrichment in plasma NEFA and TAG pools | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 4 and visit 6, following Folch extraction of the lipid moiety from plasma enrichment of 13C palmitate in NEFA and TAG pool will be measured by GCMS. The isotopic data for [13C] palmitate will be used to calculate the tracer concentration of [13C] palmitate in NEFA and TAG pool. • TAG concentration will be measured as AUC (0-240 minutes), AUC (0-360 minutes), AUC (0-480) and mean of last three points 420, 450 and 480 minutes. • The tracer concentration of [13C] palmitate in NEFA and TAG pool, will be measured as (AUC 0-240) minutes and AUC (0-480 minutes) and mean of last three points 420, 450 and 480 minutes.
[13C] 3-hydroxybutyrate enrichment relative to [13C] palmitate enrichment | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 4 and visit 6, perchloric acid treated plasma from the studies will be used to extract BOHB and the enrichment of 13C BOHB will be measured by GCMS. The isotopic data for 3-hydroxybutyrate will be used to calculate the relative partitioning of systemic plasma NEFA into [13C] 3-hydroxybutyrate as the ratio of [13C] 3-hydroxybutyrate to [13C] palmitate (in NEFA and TAG pool) in the plasma, where [13C] is expressed in micromol/L. The ratio of [13C] 3-hydroxybutyrate to [13C] palmitate (in TAG pool) in the plasma will be calculated, where [13C] is expressed in micromol/l measured as AUC (0-240 minutes), AUC (0-360 minutes), AUC (0-480 minutes) and mean of last three points 420, 450 and 480 minutes.
Glucagon, insulin and cortisol concentrations | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 4 and visit 6, the concentration of Glucagon, insulin and cortisol will be measured by RIA. Ratio of glucagon to insulin concentration will be measured as AUC (0-240 minutes), AUC (0-360 minutes), AUC (0-480) and mean of last three points 420, 450 and 480 minutes. The data will be compared following 4-weeks dapagliflozin versus placebo treatment.
Cardiac output via Transthoracic Echocardiogram | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 4 and visit 6, the cardiac output responses investigated using Echocardiogram will be compared following 4-weeks dapagliflozin versus placebo treatment.
Pulse wave velocity | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 4 and visit 6, aortic pulse wave velocity (m/s) will be measured by Vicorder between a cuff placed on the leg and around the neck. The data will be compared following 4-weeks dapagliflozin versus placebo treatment.
Plasma acylcarnitines measured by targeted metabolomics | The main analysis will be conducted once all participants have completed the metabolic studies within 2 years
  At visit 4 and visit 6, targeted metabolomics will be used to measure 188 species from the metabolome including 40 species of acyl carnitines at 480 minutes. The data will be compared following 4-weeks dapagliflozin versus placebo treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Roselle Herring, MD PhD, Principal Investigator — CEDAR, Royal Surrey County Hospital; Mellanie Davis, MD PhD, Study Chair — University of Leicester
Locations (1):
- CEDAR, Royal Surrey County Hospital, Guildford, Surrey, United Kingdom

REFERENCES:
- [Derived] Herring RA, Parsons I, Shojaee-Moradie F, Stevenage M, Jackson N, Manders R, Umpleby AM, Fielding BA, Davies M, Russell-Jones DL. Effect of Dapagliflozin on Cardiac Function and Metabolic and Hormonal Responses to Exercise. J Clin Endocrinol Metab. 2023 Mar 10;108(4):888-896. doi: 10.1210/clinem/dgac617. PMID 36274035
- [Derived] Herring RA, Shojaee-Moradie F, Stevenage M, Parsons I, Jackson N, Mendis J, Middleton B, Umpleby AM, Fielding BA, Davies M, Russell-Jones DL. The SGLT2 Inhibitor Dapagliflozin Increases the Oxidation of Ingested Fatty Acids to Ketones in Type 2 Diabetes. Diabetes Care. 2022 Jun 2;45(6):1408-1415. doi: 10.2337/dc21-2043. PMID 35312749